CLINICAL TRIAL: NCT01271933
Title: A Phase 3 Double-blind, Randomized, Placebo-controlled, Safety And Efficacy Study Of Once Daily Controlled Release Pregabalin In The Treatment Of Patients With Fibromyalgia (Protocol A0081245)
Brief Title: Study Of A Controlled Release Formulation Of Pregabalin In Fibromyalgia Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0081245; FIBROMYALGIA (Other: Alias Study Number)
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Results first posted 2018-09-14 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2018-08

CONDITIONS: Fibromyalgia
Keywords: fibromyalgia; pain; pregabalin; Lyrica
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — controlled release tablet; 165-495 mg/day; given once daily
  Arms: Pregabalin
Drug: placebo — matching placebo tablet; given once daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of a controlled release formulation of pregabalin administered once daily as compared to placebo in the treatment of fibromyalgia. All patients will receive pregabalin; half of the patients will receive placebo at some point in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have fibromyalgia.

Exclusion Criteria:

* Patients with other painful conditions cannot participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 441 (Actual)
Dates: Start 2011-03 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- United States (30):
  - Andrew O. Schreiber, MD, Orange, California
  - Apex Research Institute, Santa Ana, California
  - Paddock Park Clinical Research, Ocala, Florida
  - Broward Research Group, Pembroke Pines, Florida
  - Meridien Research, Tampa, Florida
  - Arthritis Care Center, Moline, Illinois
  - Davis Clinic, Inc, Indianapolis, Indiana
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Boston Clinical Trials, Boston, Massachusetts
  - Beacon Clinical Research, LLC, Brockton, Massachusetts
  - The Center for Pharmaceutical Research, PC, Kansas City, Missouri
  - Mercy Health Research, St Louis, Missouri
  - Quality Clinical Research, Inc., Omaha, Nebraska
  - AB Clinical Trials, Las Vegas, Nevada
  - Albuquerque Neuroscience, Incorporated, Albuquerque, New Mexico
  - Social Psychiatry Research Institute, Brooklyn, New York
  - Trinity Health Organization, Minot, North Dakota
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Radiant Research,, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - Sunstone Medical Research, LLC, Medford, Oregon
  - Allegheny Pain Management, Altoona, Pennsylvania
  - East Penn RheumatologyAssociates, P.C., Bethlehem, Pennsylvania
  - Clinical Research Associates, Inc., Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Fatigue Consultation Clinic, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Tacoma Center for Arthritis Research, PS, Tacoma, Washington
- Canada (10):
  - Dr. Alexander McIntyre Inc., Penticton, British Columbia
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Maritime Research Center, Bathurst, New Brunswick
  - Clinique Medicale Nepisiguit, Bathurst, New Brunswick
  - Tri-Hospital Sleep Laboratory West, Mississauga, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - Sleep & Alertness Research Inc., Toronto, Ontario
  - West Island Rheumatology Research Associates, Pointe-Claire, Quebec
  - Groupe de Recherche en Rhumatologie et Maladie Osseuses (GRMO Inc.), Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- India (8):
  - Mahavir Hospital & Research Centre, Hyderabad, Andhra Pradesh
  - Chanre Rheumatology & Immunology Center & Research, Bangalore, Karnataka
  - Deenanath Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Sahyadri Clinical Research & Development Center,, Pune, Maharashtra
  - Sahyadri Speciality Hospital, Pune, Maharashtra
  - Punjab Rheumatology Centre, Ludhiana, Punjab
  - Department of Rheumatology, Lucknow, Uttar Pradesh
  - Indian Spinal Injuries Centre, New Delhi
- Taiwan (4):
  - Chang Gung Medical Foundation-Linkou Branch, Kwei Shan Town, Taoyuan County
  - Chang-Hua Christian Hospital, Changhua
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei

REFERENCES:
- [Derived] Arnold LM, Arsenault P, Huffman C, Patrick JL, Messig M, Chew ML, Sanin L, Scavone JM, Pauer L, Clair AG. Once daily controlled-release pregabalin in the treatment of patients with fibromyalgia: a phase III, double-blind, randomized withdrawal, placebo-controlled study. Curr Med Res Opin. 2014 Oct;30(10):2069-83. doi: 10.1185/03007995.2014.928275. Epub 2014 Jun 27. PMID 24867298
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081245&StudyName=Study%20Of%20A%20Controlled%20Release%20Formulation%20Of%20Pregabalin%20In%20Fibromyalgia%20Patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed in 4 countries at 50 centers.
Pre-assignment Details: Baseline phase was from Visit 1 to Visit 2. Eligible participants entered single blind (SB) phase (Visit 2 to Visit 6) [6 weeks]. Responders with at least 50% improvement in pain from baseline at the end of SB phase were considered for double blind (DB) phase (Visit 6 to Visit 9) [13 weeks]. All subjects entered 1 week taper phase after completion.
Groups:
- Pregabalin (Single Blind Phase): Participants were treated with pregabalin 165 mg/day during the initial week of the SB phase.Subsequently, the pregabalin dose could have been increased based on efficacy and tolerability at each weekly visit (Visit 3 [Week 1], Visit 4 [Week 2], and Visit 5 [Week 3]).The dose could have been decreased at or between the weekly visits,up to and including Visit 5 (Week 3). The dose could only be changed by 1 step (up or down) at a time (eg, 165 mg/day to 330 mg/day, or 495 mg/day to 330 mg/day).After the end of the third week of the SB phase (Visit 5), no further dose optimization was permitted. Participants unable to tolerate a dose of at least 330 mg/day by Visit 5 (Week 3) were discontinued from the study.During the next 3 weeks of the SB phase, the optimized dose was provided. Participants unable to tolerate the optimized dose of study medication were discontinued from the study.
- Pregabalin (Double Blind Phase): At Visit 6 (Week 6), participants were randomized to receive either pregabalin at the optimized dose determined during the SB phase, or placebo. Participants randomized to pregabalin, received pregabalin at the optimized dose (330 to 495 mg/day) during the first week and thereafter. After DB baseline, all observed and volunteered AEs regardless of treatment or casually related to investigational product(s) were reported.
- Placebo (Double Blind Phase): At Visit 6 (Week 6), participants were randomized to receive either pregabalin at the optimized dose determined during the SB phase,or placebo.For participants randomized to placebo, the first week of the DB phase included a blinded taper to placebo. After DB baseline, all observed and volunteered AEs regardless of treatment or casually related to investigational product(s) were reported.
Period: Single-Blind Phase
Arm/Group | Pregabalin (Single Blind Phase) | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Started | 441 | 0 | 0
Completed | 320 | 0 | 0
Not Completed | 121 | 0 | 0
Not completed — Lack of Efficacy | 37 | 0 | 0
Not completed — Lost to Follow-up | 10 | 0 | 0
Not completed — Withdrawal by Subject | 15 | 0 | 0
Not completed — Protocol Violation | 3 | 0 | 0
Not completed — Adverse Event | 52 | 0 | 0
Not completed — (Failed to meet dosing requirement) | 1 | 0 | 0
Not completed — (Protocol non-compliance) | 2 | 0 | 0
Not completed — (Participant request-personal reason) | 1 | 0 | 0
Period: Double-Blind Phase
Arm/Group | Pregabalin (Single Blind Phase) | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Started (198 participants completed SB phase but not randomized in DB phase) | 0 | 63 | 59
Treated | 0 | 63 | 58
Completed | 0 | 46 | 47
Not Completed | 0 | 17 | 12
Not completed — Randomized but not treated | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 6 | 9
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 6 | 1
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Participant request-personal reason | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Single-blind analysis set (SBAS) consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication.
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Age, Customized [Number; unit: Participants]
  <18 years | 0
  18 - 44 years | 178
  45 - 64 years | 227
  ≥ 65 years | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 392
  Male | 49

OUTCOME MEASURES:

1. Primary Outcome: Double-Blind Phase: Time to Loss of Therapeutic Response (LTR)
Description: The time to loss of therapeutic response (LTR) is the time to loss of pain response (<30% pain response relative to the single-blind (SB) baseline mean pain) or withdrawal due to lack of efficacy or adverse events (in the double blind phase).
Time Frame: Randomization to Week 19
Population: Full analysis set (FAS) included all participants randomized to the double blind phase who received at least one dose of study medication in the double blind phase.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Days | 58 [45 to NA] — Not available was due to an insufficient number of events in a given arm to calculate the upper limit. | 23 [14 to 41]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.0186, Log Rank — The p-value was calculated using log-rank test for comparing pregabalin CR with placebo

2. Primary Outcome: Double-Blind Phase: Number of Participants With Loss of Therapeutic Response (LTR) Event
Description: Participants who did not maintain at least 30% pain response during the DB phase relative to baseline or were discontinued during DB due to lack of efficacy or an adverse event were considered to have a loss of therapeutic response.
Time Frame: Randomization to Week 19
Population: FAS included all participants randomized to the double blind phase who received at least one dose of study medication in the double blind phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Participants | 34 | 41

3. Secondary Outcome: Single-Blind Phase: Change From Baseline in Mean Daily Pain Score at Weeks 1, 2, 3, 4, 5, 6
Description: Daily Pain Score: Day 1 pain intensity over past 24 hours recorded on waking every morning. 0-10 numeric rating scale (NRS): 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  Week 1: number analyzed (Participants) | 412
  Week 1 | -0.9 (1.17)
  Week 2: number analyzed (Participants) | 409
  Week 2 | -1.5 (1.51)
  Week 3: number analyzed (Participants) | 386
  Week 3 | -2.0 (1.85)
  Week 4: number analyzed (Participants) | 363
  Week 4 | -2.3 (2.01)
  Week 5: number analyzed (Participants) | 346
  Week 5 | -2.5 (2.00)
  Week 6: number analyzed (Participants) | 330
  Week 6 | -2.6 (2.13)

4. Secondary Outcome: Double-Blind Phase: Change From Baseline in Mean Daily Pain Score at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: Daily Pain Score: Day 1 pain intensity over past 24 hours recorded on waking every morning. 0-10 NRS: 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: Full analysis set (FAS) consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Week 7: number analyzed (Participants) | 60 | 56
  Week 7 | -3.9 (1.49) | -3.0 (1.59)
  Week 8: number analyzed (Participants) | 59 | 54
  Week 8 | -3.7 (1.72) | -2.7 (1.99)
  Week 9: number analyzed (Participants) | 57 | 48
  Week 9 | -3.6 (2.01) | -2.8 (1.91)
  Week 10: number analyzed (Participants) | 57 | 49
  Week 10 | -3.7 (1.96) | -2.4 (2.01)
  Week 11: number analyzed (Participants) | 57 | 46
  Week 11 | -3.7 (2.21) | -2.6 (1.94)
  Week 12: number analyzed (Participants) | 48 | 45
  Week 12 | -3.7 (1.98) | -2.6 (1.82)
  Week 13: number analyzed (Participants) | 48 | 45
  Week 13 | -3.6 (2.10) | -2.6 (2.21)
  Week 14: number analyzed (Participants) | 48 | 43
  Week 14 | -3.5 (2.11) | -2.5 (2.14)
  Week 15: number analyzed (Participants) | 47 | 45
  Week 15 | -3.6 (2.30) | -2.6 (2.24)
  Week 16: number analyzed (Participants) | 44 | 42
  Week 16 | -3.4 (2.22) | -2.6 (1.94)
  Week 17: number analyzed (Participants) | 42 | 40
  Week 17 | -3.6 (2.02) | -2.5 (1.82)
  Week 18: number analyzed (Participants) | 42 | 41
  Week 18 | -3.4 (2.53) | -2.5 (1.93)
  Week 19: number analyzed (Participants) | 35 | 36
  Week 19 | -3.4 (2.59) | -2.4 (2.11)
  Week 20: number analyzed (Participants) | 3 | 3
  Week 20 | -3.0 (2.82) | -4.9 (2.74)

5. Secondary Outcome: Double-Blind Phase: Change From Baseline in Mean Daily Pain Score at Double Blind Endpoint Visit
Description: as for outcome 4
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase. Here, 'overall number of participants analyzed' signifies participants who were evaluable for this outcome measure.
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Units on a scale | -2.9 [-3.5 to -2.3] | -2.5 [-3.1 to -1.9]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.3310, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-1.2 to 0.4], Standard Error of Mean 0.41

6. Secondary Outcome: Single-Blind Phase: Change From Baseline in Average Daily Tiredness Score at Weeks 1, 2, 3, 4, 5, 6
Description: The tiredness assessment in the daily interactive voice response system (IVRS) diary consists of an 11-point NRS ranging from zero (not tired) to 10 (extremely tired). Participants rate their tiredness due to fibromyalgia during the past 24 hours by choosing the appropriate number between 0 (not tired) and 10 (extremely tired).
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: SBAS consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  Week 1: number analyzed (Participants) | 412
  Week 1 | -0.7 (1.16)
  Week 2: number analyzed (Participants) | 409
  Week 2 | -1.2 (1.53)
  Week 3: number analyzed (Participants) | 386
  Week 3 | -1.6 (1.91)
  Week 4: number analyzed (Participants) | 362
  Week 4 | -2.0 (2.08)
  Week 5: number analyzed (Participants) | 346
  Week 5 | -2.2 (2.10)
  Week 6: number analyzed (Participants) | 331
  Week 6 | -2.3 (2.17)

7. Secondary Outcome: Double-Blind Phase: Change From Baseline in Average Daily Tiredness Score at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: The tiredness assessment in the daily IVRS diary consists of an 11-point NRS ranging from zero (not tired) to 10 (extremely tired). Participants rate their tiredness due to fibromyalgia during the past 24 hours by choosing the appropriate number between 0 (not tired) and 10 (extremely tired).
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Week 7: number analyzed (Participants) | 60 | 56
  Week 7 | -3.4 (1.74) | -3.0 (1.79)
  Week 8: number analyzed (Participants) | 59 | 54
  Week 8 | -3.3 (1.81) | -2.8 (1.95)
  Week 9: number analyzed (Participants) | 57 | 48
  Week 9 | -3.2 (1.93) | -2.9 (1.98)
  Week 10: number analyzed (Participants) | 57 | 49
  Week 10 | -3.2 (2.03) | -2.6 (1.93)
  Week 11: number analyzed (Participants) | 57 | 46
  Week 11 | -3.1 (2.16) | -2.5 (1.91)
  Week 12: number analyzed (Participants) | 48 | 45
  Week 12 | -3.4 (1.77) | -2.5 (1.69)
  Week 13: number analyzed (Participants) | 48 | 45
  Week 13 | -3.2 (1.82) | -2.6 (1.87)
  Week 14: number analyzed (Participants) | 48 | 43
  Week 14 | -3.2 (2.06) | -2.5 (1.95)
  Week 15: number analyzed (Participants) | 47 | 45
  Week 15 | -3.4 (2.15) | -2.6 (1.96)
  Week 16: number analyzed (Participants) | 44 | 42
  Week 16 | -3.1 (2.15) | -2.7 (1.84)
  Week 17: number analyzed (Participants) | 42 | 40
  Week 17 | -3.4 (1.88) | -2.5 (1.96)
  Week 18: number analyzed (Participants) | 42 | 41
  Week 18 | -3.2 (2.24) | -2.4 (1.82)
  Week 19: number analyzed (Participants) | 35 | 36
  Week 19 | -3.1 (2.23) | -2.4 (1.96)
  Week 20: number analyzed (Participants) | 3 | 3
  Week 20 | -2.7 (2.42) | -4.9 (1.48)

8. Secondary Outcome: Double-Blind Phase: Change From Baseline in Average Daily Tiredness Score at Double Blind Endpoint Visit
Description: as for outcome 7
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Units on a scale | -2.6 [-3.2 to -2.0] | -2.5 [-3.1 to -1.9]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.9247, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-0.8 to 0.8], Standard Error of Mean 0.40

9. Secondary Outcome: Single-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Wake After Sleep and Subjective Latency to Sleep Onset at Weeks 1, 2, 3, 4, 5, 6
Description: The SSQ is designed to capture subjective behavior in participants with disrupted sleep. Participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (NRS) for the previous night.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Minutes
  Subjective Wake after Sleep Onset (Week 1): number analyzed (Participants) | 410
  Subjective Wake after Sleep Onset (Week 1) | -19.1 (45.90)
  Subjective Wake after Sleep Onset (Week 2): number analyzed (Participants) | 405
  Subjective Wake after Sleep Onset (Week 2) | -22.4 (50.22)
  Subjective Wake after Sleep Onset (Week 3): number analyzed (Participants) | 384
  Subjective Wake after Sleep Onset (Week 3) | -25.0 (64.57)
  Subjective Wake after Sleep Onset (Week 4): number analyzed (Participants) | 360
  Subjective Wake after Sleep Onset (Week 4) | -27.5 (62.58)
  Subjective Wake after Sleep Onset (Week 5): number analyzed (Participants) | 346
  Subjective Wake after Sleep Onset (Week 5) | -31.4 (57.37)
  Subjective Wake after Sleep Onset (Week 6): number analyzed (Participants) | 331
  Subjective Wake after Sleep Onset (Week 6) | -32.8 (59.51)
  Subjective Latency to Sleep Onset (Week 1): number analyzed (Participants) | 412
  Subjective Latency to Sleep Onset (Week 1) | -10.3 (42.35)
  Subjective Latency to Sleep Onset (Week 2): number analyzed (Participants) | 409
  Subjective Latency to Sleep Onset (Week 2) | -13.0 (43.25)
  Subjective Latency to Sleep Onset (Week 3): number analyzed (Participants) | 386
  Subjective Latency to Sleep Onset (Week 3) | -15.5 (49.01)
  Subjective Latency to Sleep Onset (Week 4): number analyzed (Participants) | 362
  Subjective Latency to Sleep Onset (Week 4) | -19.6 (49.84)
  Subjective Latency to Sleep Onset (Week 5): number analyzed (Participants) | 346
  Subjective Latency to Sleep Onset (Week 5) | -20.0 (52.32)
  Subjective Latency to Sleep Onset (Week 6): number analyzed (Participants) | 331
  Subjective Latency to Sleep Onset (Week 6) | -16.9 (47.34)

10. Secondary Outcome: Single-Blind Phase: Change From Baseline in Daily SSQ - Subjective Number of Awakenings After Sleep Onset at Weeks 1, 2, 3, 4, 5, 6
Description: as for outcome 9
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: SBAS consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication. Here, 'overall number of participants analyzed' signifies participants who awakened after sleep.
Measure: Mean (Standard Deviation); unit: Number of times the participant awakened
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 439
Number of times the participant awakened
  Subjective No.of Awakenings after Sleep (Week 1): number analyzed (Participants) | 410
  Subjective No.of Awakenings after Sleep (Week 1) | -0.8 (1.28)
  Subjective No.of Awakenings after Sleep (Week 2): number analyzed (Participants) | 405
  Subjective No.of Awakenings after Sleep (Week 2) | -1.0 (1.50)
  Subjective No.of Awakenings after Sleep (Week 3): number analyzed (Participants) | 384
  Subjective No.of Awakenings after Sleep (Week 3) | -1.1 (1.54)
  Subjective No.of Awakenings after Sleep (Week 4): number analyzed (Participants) | 360
  Subjective No.of Awakenings after Sleep (Week 4) | -1.1 (1.44)
  Subjective No.of Awakenings after Sleep (Week 5): number analyzed (Participants) | 346
  Subjective No.of Awakenings after Sleep (Week 5) | -1.2 (1.70)
  Subjective No.of Awakenings after Sleep (Week 6): number analyzed (Participants) | 331
  Subjective No.of Awakenings after Sleep (Week 6) | -1.2 (1.52)

11. Secondary Outcome: Single-Blind Phase: Change From Baseline in Daily SSQ - Subjective Total Sleep Time at Weeks 1, 2, 3, 4, 5, 6
Description: as for outcome 9
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Hours
  Subjective Total Sleep Time (Week 1): number analyzed (Participants) | 411
  Subjective Total Sleep Time (Week 1) | 0.6 (0.93)
  Subjective Total Sleep Time (Week 2): number analyzed (Participants) | 407
  Subjective Total Sleep Time (Week 2) | 0.6 (0.96)
  Subjective Total Sleep Time (Week 3): number analyzed (Participants) | 385
  Subjective Total Sleep Time (Week 3) | 0.6 (1.00)
  Subjective Total Sleep Time (Week 4): number analyzed (Participants) | 360
  Subjective Total Sleep Time (Week 4) | 0.7 (0.94)
  Subjective Total Sleep Time (Week 5): number analyzed (Participants) | 346
  Subjective Total Sleep Time (Week 5) | 0.7 (1.00)
  Subjective Total Sleep Time (Week 6): number analyzed (Participants) | 331
  Subjective Total Sleep Time (Week 6) | 0.7 (1.08)

12. Secondary Outcome: Single-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Sleep Quality at Weeks 1, 2, 3, 4, 5, 6
Description: The SSQ is designed to capture subjective behavior in participants with disrupted sleep. Participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (NRS) for the previous night. Participants rated quality of sleep during the past night by selecting a number between 0 (very poor) and 10 (excellent). Mean sleep quality was calculated as the mean of the last seven days, the potential range of responses at each week was therefore 0 (very poor) -10 (excellent), where higher scores indicated better quality of sleep.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 5, 6
Population: SBAS consisted of all participants who were enrolled into the SB phase of the study and received at least 1 dose of study medication. Here, 'overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 439
Units on a scale
  Sleep quality (Week 1): number analyzed (Participants) | 410
  Sleep quality (Week 1) | 1.0 (1.35)
  Sleep quality (Week 2): number analyzed (Participants) | 405
  Sleep quality (Week 2) | 1.2 (1.43)
  Sleep quality (Week 3): number analyzed (Participants) | 384
  Sleep quality (Week 3) | 1.5 (1.75)
  Sleep quality (Week 4): number analyzed (Participants) | 360
  Sleep quality (Week 4) | 1.6 (1.79)
  Sleep quality (Week 5): number analyzed (Participants) | 346
  Sleep quality (Week 5) | 1.7 (1.82)
  Sleep quality (Week 6): number analyzed (Participants) | 330
  Sleep quality (Week 6) | 1.7 (1.89)

13. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Wake After Sleep Onset and Subjective Latency to Sleep Onset at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: as for outcome 9
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Minutes
  Subjective Wake after Sleep Onset (Week 7): number analyzed (Participants) | 60 | 56
  Subjective Wake after Sleep Onset (Week 7) | -27.8 (37.29) | -32.0 (50.47)
  Subjective Wake after Sleep Onset (Week 8): number analyzed (Participants) | 59 | 54
  Subjective Wake after Sleep Onset (Week 8) | -27.4 (39.39) | -28.0 (56.99)
  Subjective Wake after Sleep Onset (Week 9): number analyzed (Participants) | 57 | 48
  Subjective Wake after Sleep Onset (Week 9) | -27.0 (40.12) | -33.2 (56.45)
  Subjective Wake after Sleep Onset (Week 10): number analyzed (Participants) | 57 | 49
  Subjective Wake after Sleep Onset (Week 10) | -26.9 (38.92) | -26.2 (68.24)
  Subjective Wake after Sleep Onset (Week 11): number analyzed (Participants) | 57 | 46
  Subjective Wake after Sleep Onset (Week 11) | -29.0 (44.80) | -37.4 (56.79)
  Subjective Wake after Sleep Onset (Week 12): number analyzed (Participants) | 48 | 45
  Subjective Wake after Sleep Onset (Week 12) | -26.0 (46.00) | -31.0 (43.96)
  Subjective Wake after Sleep Onset (Week 13): number analyzed (Participants) | 48 | 44
  Subjective Wake after Sleep Onset (Week 13) | -22.8 (37.78) | -31.4 (50.08)
  Subjective Wake after Sleep Onset (Week 14): number analyzed (Participants) | 48 | 43
  Subjective Wake after Sleep Onset (Week 14) | -27.0 (39.87) | -43.3 (54.45)
  Subjective Wake after Sleep Onset (Week 15): number analyzed (Participants) | 47 | 45
  Subjective Wake after Sleep Onset (Week 15) | -31.7 (38.37) | -35.1 (56.47)
  Subjective Wake after Sleep Onset (Week 16): number analyzed (Participants) | 43 | 42
  Subjective Wake after Sleep Onset (Week 16) | -25.9 (41.95) | -35.0 (52.67)
  Subjective Wake after Sleep Onset (Week 17): number analyzed (Participants) | 42 | 40
  Subjective Wake after Sleep Onset (Week 17) | -31.5 (34.29) | -36.2 (58.67)
  Subjective Wake after Sleep Onset (Week 18): number analyzed (Participants) | 42 | 40
  Subjective Wake after Sleep Onset (Week 18) | -32.4 (36.37) | -37.3 (56.67)
  Subjective Wake after Sleep Onset (Week 19): number analyzed (Participants) | 35 | 36
  Subjective Wake after Sleep Onset (Week 19) | -27.3 (52.27) | -23.1 (46.28)
  Subjective Wake after Sleep Onset (Week 20): number analyzed (Participants) | 3 | 3
  Subjective Wake after Sleep Onset (Week 20) | -22.5 (11.03) | -7.1 (11.15)
  Subjective Latency to Sleep Onset (Week 7): number analyzed (Participants) | 60 | 56
  Subjective Latency to Sleep Onset (Week 7) | -15.6 (55.67) | -19.1 (41.02)
  Subjective Latency to Sleep Onset (Week 8): number analyzed (Participants) | 59 | 54
  Subjective Latency to Sleep Onset (Week 8) | -19.1 (29.70) | -12.3 (42.83)
  Subjective Latency to Sleep Onset (Week 9): number analyzed (Participants) | 57 | 48
  Subjective Latency to Sleep Onset (Week 9) | -18.4 (34.03) | -16.0 (50.97)
  Subjective Latency to Sleep Onset (Week 10): number analyzed (Participants) | 57 | 49
  Subjective Latency to Sleep Onset (Week 10) | -19.5 (29.40) | -18.0 (43.83)
  Latency to Sleep Onset (Week 11): number analyzed (Participants) | 57 | 46
  Latency to Sleep Onset (Week 11) | -18.5 (22.40) | -18.0 (47.82)
  Subjective Latency to Sleep Onset (Week 12): number analyzed (Participants) | 48 | 45
  Subjective Latency to Sleep Onset (Week 12) | -16.3 (26.04) | -18.8 (40.31)
  Subjective Latency to Sleep Onset (Week 13): number analyzed (Participants) | 48 | 44
  Subjective Latency to Sleep Onset (Week 13) | -17.5 (20.79) | -16.8 (36.51)
  Subjective Latency to Sleep Onset (Week 14): number analyzed (Participants) | 48 | 43
  Subjective Latency to Sleep Onset (Week 14) | -20.8 (25.58) | -21.8 (44.03)
  Subjective Latency to Sleep Onset (Week 15): number analyzed (Participants) | 47 | 45
  Subjective Latency to Sleep Onset (Week 15) | -19.4 (20.25) | -19.1 (42.55)
  Subjective Latency to Sleep Onset (Week 16): number analyzed (Participants) | 44 | 42
  Subjective Latency to Sleep Onset (Week 16) | -15.8 (31.85) | -20.9 (42.18)
  Subjective Latency to Sleep Onset (Week 17): number analyzed (Participants) | 42 | 40
  Subjective Latency to Sleep Onset (Week 17) | -23.1 (23.09) | -20.9 (49.30)
  Subjective Latency to Sleep Onset (Week 18): number analyzed (Participants) | 42 | 40
  Subjective Latency to Sleep Onset (Week 18) | -16.3 (24.52) | -18.7 (46.23)
  Subjective Latency to Sleep Onset (Week 19): number analyzed (Participants) | 35 | 36
  Subjective Latency to Sleep Onset (Week 19) | -16.7 (29.38) | -19.5 (50.89)
  Subjective Latency to Sleep Onset (Week 20): number analyzed (Participants) | 3 | 3
  Subjective Latency to Sleep Onset (Week 20) | 23.0 (84.31) | -28.7 (8.00)

14. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Number of Awakenings After Sleep Onset at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: as for outcome 9
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Number of times the participant awakened
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Number of times the participant awakened
  Subjective No.of Awakenings after Sleep (Week 7): number analyzed (Participants) | 60 | 56
  Subjective No.of Awakenings after Sleep (Week 7) | -1.1 (1.39) | -1.0 (1.30)
  Subjective No.of Awakenings after Sleep (Week 8): number analyzed (Participants) | 59 | 54
  Subjective No.of Awakenings after Sleep (Week 8) | -1.2 (1.23) | -0.8 (1.27)
  Subjective No.of Awakenings after Sleep (Week 9): number analyzed (Participants) | 57 | 48
  Subjective No.of Awakenings after Sleep (Week 9) | -1.2 (0.94) | -1.1 (1.12)
  Subjective No.of Awakenings after Sleep (Week 10): number analyzed (Participants) | 57 | 49
  Subjective No.of Awakenings after Sleep (Week 10) | -1.2 (1.10) | -0.9 (1.16)
  Subjective No.of Awakenings after Sleep (Week 11): number analyzed (Participants) | 57 | 46
  Subjective No.of Awakenings after Sleep (Week 11) | -1.1 (1.40) | -0.9 (1.18)
  Subjective No.of Awakenings after Sleep (Week 12): number analyzed (Participants) | 48 | 45
  Subjective No.of Awakenings after Sleep (Week 12) | -1.1 (1.50) | -0.8 (1.00)
  Subjective No.of Awakenings after Sleep (Week 13): number analyzed (Participants) | 48 | 44
  Subjective No.of Awakenings after Sleep (Week 13) | -1.0 (1.02) | -1.0 (1.13)
  Subjective No.of Awakenings after Sleep (Week 14): number analyzed (Participants) | 48 | 43
  Subjective No.of Awakenings after Sleep (Week 14) | -1.0 (1.06) | -1.1 (1.07)
  Subjective No.of Awakenings after Sleep (Week 15): number analyzed (Participants) | 47 | 45
  Subjective No.of Awakenings after Sleep (Week 15) | -0.8 (2.20) | -1.1 (1.21)
  Subjective No.of Awakenings after Sleep (Week 16): number analyzed (Participants) | 43 | 42
  Subjective No.of Awakenings after Sleep (Week 16) | -1.0 (1.10) | -1.0 (1.18)
  Subjective No.of Awakenings after Sleep (Week 17): number analyzed (Participants) | 42 | 40
  Subjective No.of Awakenings after Sleep (Week 17) | -1.2 (0.92) | -0.9 (1.25)
  Subjective No.of Awakenings after Sleep (Week 18): number analyzed (Participants) | 42 | 40
  Subjective No.of Awakenings after Sleep (Week 18) | -1.1 (1.14) | -1.0 (1.28)
  Subjective No.of Awakenings after Sleep (Week 19): number analyzed (Participants) | 35 | 36
  Subjective No.of Awakenings after Sleep (Week 19) | -0.7 (2.63) | -0.9 (1.32)
  Subjective No.of Awakenings after Sleep (Week 20): number analyzed (Participants) | 3 | 3
  Subjective No.of Awakenings after Sleep (Week 20) | -1.5 (1.14) | -1.5 (0.95)

15. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Total Sleep Time at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: The SSQ is designed to capture subjective behavior in participants with disrupted sleep. Participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (NRS) for the previous night. Subjective total sleep time was the subjective estimate of the total amount of time the participant was asleep after lights out until final awakening.
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Hours
  Subjective Total Sleep Time (Week 7): number analyzed (Participants) | 60 | 56
  Subjective Total Sleep Time (Week 7) | 0.7 (1.00) | 0.5 (1.10)
  Subjective Total Sleep Time (Week 8): number analyzed (Participants) | 59 | 54
  Subjective Total Sleep Time (Week 8) | 0.9 (0.89) | 0.6 (1.25)
  Subjective Total Sleep Time (Week 9): number analyzed (Participants) | 57 | 48
  Subjective Total Sleep Time (Week 9) | 0.8 (1.00) | 0.5 (1.10)
  Subjective Total Sleep Time (Week 10): number analyzed (Participants) | 57 | 49
  Subjective Total Sleep Time (Week 10) | 0.9 (1.07) | 0.5 (1.01)
  Subjective Total Sleep Time (Week 11): number analyzed (Participants) | 57 | 46
  Subjective Total Sleep Time (Week 11) | 0.9 (0.86) | 0.6 (1.08)
  Subjective Total Sleep Time (Week 12): number analyzed (Participants) | 48 | 45
  Subjective Total Sleep Time (Week 12) | 0.8 (1.01) | 0.5 (1.13)
  Subjective Total Sleep Time (Week 13): number analyzed (Participants) | 48 | 44
  Subjective Total Sleep Time (Week 13) | 0.7 (0.93) | 0.6 (0.95)
  Subjective Total Sleep Time (Week 14): number analyzed (Participants) | 48 | 43
  Subjective Total Sleep Time (Week 14) | 0.9 (1.31) | 0.7 (1.17)
  Subjective Total Sleep Time (Week 15): number analyzed (Participants) | 47 | 45
  Subjective Total Sleep Time (Week 15) | 0.7 (0.90) | 0.7 (1.22)
  Subjective Total Sleep Time (Week 16): number analyzed (Participants) | 44 | 42
  Subjective Total Sleep Time (Week 16) | 0.7 (0.94) | 0.7 (1.04)
  Subjective Total Sleep Time (Week 17): number analyzed (Participants) | 42 | 40
  Subjective Total Sleep Time (Week 17) | 0.7 (0.85) | 0.7 (1.08)
  Subjective Total Sleep Time (Week 18): number analyzed (Participants) | 42 | 40
  Subjective Total Sleep Time (Week 18) | 0.6 (0.85) | 0.5 (1.23)
  Subjective Total Sleep Time (Week 19): number analyzed (Participants) | 35 | 36
  Subjective Total Sleep Time (Week 19) | 0.5 (1.10) | 0.6 (1.15)
  Subjective Total Sleep Time (Week 20): number analyzed (Participants) | 3 | 3
  Subjective Total Sleep Time (Week 20) | -0.1 (1.02) | 0.5 (0.41)

16. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Sleep Quality at Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Description: as for outcome 12
Time Frame: Baseline, Weeks 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Sleep Quality (Week 7): number analyzed (Participants) | 60 | 56
  Sleep Quality (Week 7) | 1.9 (1.69) | 1.9 (1.62)
  Sleep Quality (Week 8): number analyzed (Participants) | 59 | 53
  Sleep Quality (Week 8) | 2.0 (1.61) | 1.7 (1.71)
  Sleep Quality (Week 9): number analyzed (Participants) | 57 | 48
  Sleep Quality (Week 9) | 2.1 (1.47) | 1.8 (1.66)
  Sleep Quality (Week 10): number analyzed (Participants) | 57 | 49
  Sleep Quality (Week 10) | 2.2 (1.70) | 1.7 (1.74)
  Sleep Quality (Week 11): number analyzed (Participants) | 57 | 46
  Sleep Quality (Week 11) | 2.3 (1.78) | 1.7 (1.63)
  Sleep Quality (Week 12): number analyzed (Participants) | 48 | 45
  Sleep Quality (Week 12) | 2.1 (1.66) | 1.7 (1.65)
  Sleep Quality (Week 13): number analyzed (Participants) | 48 | 44
  Sleep Quality (Week 13) | 1.9 (1.72) | 1.9 (1.63)
  Sleep Quality (Week 14) N=48,43: number analyzed (Participants) | 48 | 43
  Sleep Quality (Week 14) N=48,43 | 2.2 (1.69) | 2.1 (1.73)
  Sleep Quality (Week 15): number analyzed (Participants) | 47 | 45
  Sleep Quality (Week 15) | 2.2 (1.76) | 2.0 (1.64)
  Sleep Quality (Week 16): number analyzed (Participants) | 43 | 42
  Sleep Quality (Week 16) | 1.9 (1.87) | 1.9 (1.68)
  Sleep Quality (Week 17): number analyzed (Participants) | 42 | 40
  Sleep Quality (Week 17) | 2.2 (1.71) | 1.9 (1.72)
  Sleep Quality (Week 18): number analyzed (Participants) | 42 | 40
  Sleep Quality (Week 18) | 2.1 (1.64) | 1.8 (1.71)
  Sleep Quality (Week 19): number analyzed (Participants) | 35 | 36
  Sleep Quality (Week 19) | 2.0 (1.77) | 1.5 (1.55)
  Sleep Quality (Week 20): number analyzed (Participants) | 3 | 3
  Sleep Quality (Week 20) | 3.1 (1.23) | 3.3 (0.45)

17. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Wake After Sleep Onset and Subjective Latency to Sleep Onset at Double Blind Endpoint Visit
Description: as for outcome 9
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Minutes
  Subjective Wake after Sleep Onset | -26.2 [-36.6 to -15.8] | -20.6 [-30.7 to -10.5]
  Subjective Latency to Sleep Onset | -10.6 [-24.2 to 3.0] | -11.9 [-25.0 to 1.3]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Subjective Wake after Sleep Onset; Test type: Superiority or Other; p = 0.4314, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -5.6, 95% CI 2-sided [-19.7 to 8.5], Standard Error of Mean 7.12
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Subjective Latency to Sleep Onset; Test type: Superiority or Other; p = 0.8915, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-17.1 to 19.6], Standard Error of Mean 9.26

18. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Number of Awakenings After Sleep Onset at Double Blind Endpoint Visit
Description: as for outcome 9
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Number of times the participant awakened
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Number of times the participant awakened | -0.5 [-1.1 to 0.1] | -0.8 [-1.4 to -0.2]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.4571, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.1], Standard Error of Mean 0.41

19. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Subjective Total Sleep Time at Double Blind Endpoint Visit
Description: as for outcome 9
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Hours | 0.6 [0.3 to 0.9] | 0.4 [0.1 to 0.7]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.3779, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.20

20. Secondary Outcome: Double-Blind Phase: Change From Baseline in Daily Subjective Sleep Questionnaire (SSQ) - Sleep Quality at Double Blind Endpoint Visit
Description: The SSQ is designed to capture subjective behavior in participants with disrupted sleep. Participants report latency (how long it took them to fall asleep), how many hours they slept, the number of times they woke up, the total wake time after sleep onset, and then rate the quality of their sleep (NRS) for the previous night. Participants rated quality of sleep during the past night by selecting a number between 0 (very poor) and 10 (excellent).
Time Frame: Baseline, Double blind endpoint visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 62 | 58
Units on a scale | 1.9 [1.4 to 2.4] | 1.4 [1.0 to 1.9]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.2009, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.2 to 1.1], Standard Error of Mean 0.34

21. Secondary Outcome: Single-Blind Phase: Change From Baseline in Weekly Pain Score at Week 6 (1 Week Recall Period)
Description: Weekly pain scores were calculated from the daily pain diary. Daily Pain Score: Day 1 pain intensity over past 24 hours recorded on waking every morning. 0-10 NRS: 0 (no pain) to 10 (worst possible pain).
Time Frame: Baseline, Week 6
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 289
Units on a scale | -1.6 (2.18)

22. Secondary Outcome: Double-Blind Phase: Change From Baseline in Weekly Pain Score at Week 19 (1 Week Recall Period)
Description: as for outcome 21
Time Frame: Baseline, Week 19
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 60 | 57
Units on a scale | -3.1 [-3.8 to -2.4] | -2.4 [-3.1 to -1.7]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.1845, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-1.6 to 0.3], Standard Error of Mean 0.48

23. Secondary Outcome: Change From Baseline in Medical Outcomes Study-Sleep Scale (MOS-SS) at Week 6 - Sleep Disturbance, Snoring, Awakening Short of Breath or With a Headache, Sleep Adequacy, Somnolence, Sleep Problems Index I and Sleep Problems Index II
Description: The MOS-SS is a validated self-administered questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) and two overall sleep problems indices assessing sleep over the past week. Score range for Sleep Disturbance (SD), sleep adequacy (SA), snoring, somnolence, awakening short of breath/headache was 0-100, where higher score=greater SD; greater SA; greater snoring; greater somnolence; greater shortness of breath/headache respectively. Quantity of Sleep (range-0 to 24 hours; higher scores/hours=greater quantity of sleep). Sleep Problem Index I and II: Score Range=0 to 100; higher scores =greater sleep problems. Optimal Sleep (assessed as yes or no), 'Yes' =optimal sleep (average 7-8 hours/night); 'No' =not optimal sleep.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  Sleep disturbance: number analyzed (Participants) | 289
  Sleep disturbance | -21.8 (24.82)
  Snoring: number analyzed (Participants) | 281
  Snoring | -1.0 (24.94)
  Awakening Short of Breath/with a Headache: number analyzed (Participants) | 288
  Awakening Short of Breath/with a Headache | -11.0 (30.59)
  Sleep adequacy: number analyzed (Participants) | 289
  Sleep adequacy | 18.9 (31.17)
  Somnolence: number analyzed (Participants) | 289
  Somnolence | -3.6 (24.87)
  Sleep Problems Index I: number analyzed (Participants) | 288
  Sleep Problems Index I | -16.1 (21.62)
  Sleep Problems Index II: number analyzed (Participants) | 288
  Sleep Problems Index II | -15.9 (20.44)

24. Secondary Outcome: Change From Baseline in Medical Outcomes Study-Sleep Scale (MOS-SS) at Week 6- Quantity of Sleep
Description: as for outcome 23
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
hours | 0.7 (1.33)

25. Secondary Outcome: Double-Blind Phase: Change From Baseline in Medical Outcomes Study-Sleep Scale (MOS-SS) at Week 19-Sleep Disturbance, Snoring, Awakening Short of Breath or With a Headache, Sleep Adequacy, Somnolence, Sleep Problems Index I and Sleep Problems Index II
Description: as for outcome 23
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Sleep disturbance: number analyzed (Participants) | 60 | 57
  Sleep disturbance | -25.4 [-32.0 to -18.8] | -15.5 [-21.8 to -9.1]
  Snoring: number analyzed (Participants) | 58 | 56
  Snoring | -2.4 [-5.2 to 9.9] | -2.9 [-10.1 to 4.3]
  Awakening Short of Breath/with a Headache: number analyzed (Participants) | 59 | 57
  Awakening Short of Breath/with a Headache | -8.1 [-13.5 to -2.7] | -4.2 [-9.3 to -0.9]
  Sleep adequacy: number analyzed (Participants) | 60 | 57
  Sleep adequacy | 23.9 [16.0 to 31.9] | 17.1 [9.5 to 24.8]
  Somnolence: number analyzed (Participants) | 60 | 57
  Somnolence | -11.9 [-17.8 to -5.9] | -6.6 [-12.4 to -0.9]
  Sleep Problems Index I: number analyzed (Participants) | 59 | 57
  Sleep Problems Index I | -19.5 [-25.0 to -13.9] | -13.7 [-19.0 to -8.3]
  Sleep Problems Index II: number analyzed (Participants) | 59 | 57
  Sleep Problems Index II | -19.7 [-25.4 to -14.0] | -14.0 [-19.5 to -8.6]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Sleep disturbance; Test type: Superiority or Other; p = 0.0305, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-18.9 to 1.0], Standard Error of Mean 4.52
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Snoring; Test type: Superiority or Other; p = 0.3133, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [-5.0 to 15.5], Standard Error of Mean 5.17
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Awakening Short of Breath or with a Headache; Test type: Superiority or Other; p = 0.2985, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-11.2 to 3.5], Standard Error of Mean 3.71
Statistical Analysis 4: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Sleep adequacy; Test type: Superiority or Other; p = 0.2159, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 6.8, 95% CI 2-sided [-4.1 to 17.7], Standard Error of Mean 5.49
Statistical Analysis 5: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Somnolence; Test type: Superiority or Other; p = 0.2041, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -5.2, 95% CI 2-sided [-13.4 to 2.9], Standard Error of Mean 4.10
Statistical Analysis 6: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Sleep Problems Index I; Test type: Superiority or Other; p = 0.1319, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -5.8, 95% CI 2-sided [-13.4 to 1.8], Standard Error of Mean 3.81
Statistical Analysis 7: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Sleep Problems Index II; Test type: Superiority or Other; p = 0.1473, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -5.7, 95% CI 2-sided [-13.4 to 2.0], Standard Error of Mean 3.89

26. Secondary Outcome: Double-Blind Phase: Change From Baseline in Medical Outcomes Study-Sleep Scale (MOS-SS) at Week 19- Quantity of Sleep
Description: as for outcome 23
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: hours
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
hours | 0.7 [0.4 to 1.0] | 0.5 [0.2 to 0.8]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.3596, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.6], Standard Error of Mean 0.20

27. Secondary Outcome: Single-Blind Phase: Number of Participants Who Reported Global Impression of Change (PGIC) at Week 6
Description: PGIC: participant rated instrument to measure participant's change in overall status on a 7-point scale; range from 1 (very much improved) to 7 (very much worse).
Time Frame: Week 6
Population: as for outcome 12
Measure: Number; unit: Participants
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 289
Participants
  Very Much Improved | 24
  Much Improved | 77
  Minimally Improved | 103
  No Change | 46
  Minimally Worse | 16
  Much Worse | 18
  Very Much Worse | 5

28. Secondary Outcome: Double-Blind Phase: Number of Participants Who Reported Global Impression of Change (PGIC) at Week 19
Description: as for outcome 27
Time Frame: Week 19
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 60 | 57
Participants
  Very Much Improved | 7 | 7
  Much Improved | 15 | 11
  Minimally Improved | 14 | 12
  No Change | 9 | 11
  Minimally Worse | 7 | 6
  Much Worse | 7 | 8
  Very Much Worse | 1 | 2
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Odds ratio is the probability of the event occurring in Pregabalin 330 - 495 mg/day relative to the event occurring in Placebo for Pregabalin. Odds ratio > 1 is in favor of Pregabalin 330 - 495 mg/day; Test type: Superiority or Other; p = 0.4985, two-sided test — Nominal p-value for two-sided test; Odds Ratio (OR) = 1.25, 95% CI 2-sided [0.66 to 2.36]

29. Secondary Outcome: Single-Blind Phase: Change From Baseline in 36-Item Short-Form Health Survey (SF-36) at Week 6
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, mental health. The score for a section is an average of the individual question scores, which are scaled 0-100. Higher scores indicated a better health-related quality of life.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  SF-36 Physical Functioning: number analyzed (Participants) | 420
  SF-36 Physical Functioning | 14.0 (19.89)
  SF-36 Role-Physical: number analyzed (Participants) | 420
  SF-36 Role-Physical | 17.8 (27.38)
  SF-36 Pain Index: number analyzed (Participants) | 420
  SF-36 Pain Index | 20.7 (22.07)
  SF-36 General Health Perceptions: number analyzed (Participants) | 420
  SF-36 General Health Perceptions | 8.5 (17.96)
  SF-36 Vitality: number analyzed (Participants) | 420
  SF-36 Vitality | 18.2 (24.35)
  SF-36 Social Functioning: number analyzed (Participants) | 420
  SF-36 Social Functioning | 12.9 (28.19)
  SF-36 Role-Emotional: number analyzed (Participants) | 420
  SF-36 Role-Emotional | 8.6 (29.40)
  SF-36 Mental Health Index: number analyzed (Participants) | 420
  SF-36 Mental Health Index | 7.9 (18.94)
  Physical Component Score: number analyzed (Participants) | 420
  Physical Component Score | 7.2 (8.75)
  Mental Component Score: number analyzed (Participants) | 420
  Mental Component Score | 4.5 (11.78)

30. Secondary Outcome: Double-Blind Phase: Change From Baseline in SF-36 Score at Week 19
Description: as for outcome 29
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  SF-36 Physical Functioning: number analyzed (Participants) | 60 | 57
  SF-36 Physical Functioning | 12.4 [6.4 to 18.4] | 13.7 [8.0 to 19.5]
  SF-36 Role-Physical: number analyzed (Participants) | 60 | 57
  SF-36 Role-Physical | 18.9 [11.7 to 26.0] | 16.2 [9.4 to 23.1]
  SF-36 Pain Index: number analyzed (Participants) | 60 | 57
  SF-36 Pain Index | 19.2 [12.5 to 26.0] | 16.0 [9.5 to 22.5]
  SF-36 General Health Perceptions: number analyzed (Participants) | 60 | 57
  SF-36 General Health Perceptions | 3.3 [-1.8 to 8.3] | 9.3 [4.5 to 14.2]
  SF-36 Vitality: number analyzed (Participants) | 60 | 57
  SF-36 Vitality | 12.2 [5.3 to 19.1] | 15.7 [9.1 to 22.3]
  SF-36 Social Functioning: number analyzed (Participants) | 60 | 57
  SF-36 Social Functioning | 13.3 [7.0 to 19.6] | 13.5 [7.4 to 19.5]
  SF-36 Role-Emotional: number analyzed (Participants) | 60 | 57
  SF-36 Role-Emotional | 3.8 [-4.1 to 11.7] | 2.2 [-5.4 to 9.8]
  SF-36 Mental Health Index: number analyzed (Participants) | 60 | 57
  SF-36 Mental Health Index | 6.6 [1.4 to 11.7] | 5.2 [0.3 to 10.2]
  Physical Component Score: number analyzed (Participants) | 60 | 57
  Physical Component Score | 6.8 [4.2 to 9.4] | 7.2 [4.7 to 9.7]
  Mental Component Score: number analyzed (Participants) | 60 | 57
  Mental Component Score | 2.6 [-0.6 to 5.8] | 2.4 [-0.7 to 5.5]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Physical Functioning; Test type: Superiority or Other; p = 0.7400, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-9.5 to 6.8], Standard Error of Mean 4.10
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Role-Physical; Test type: Superiority or Other; p = 0.5938, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [-7.1 to 12.3], Standard Error of Mean 4.89
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Pain Index; Test type: Superiority or Other; p = 0.4842, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-5.9 to 12.4], Standard Error of Mean 4.61
Statistical Analysis 4: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 General Health Perceptions; Test type: Superiority or Other; p = 0.0827, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -6.1, 95% CI 2-sided [-12.9 to 0.8], Standard Error of Mean 3.45
Statistical Analysis 5: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Vitality; Test type: Superiority or Other; p = 0.4561, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-12.09 to 5.8], Standard Error of Mean 4.73
Statistical Analysis 6: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Social Functioning; Test type: Superiority or Other; p = 0.9645, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-8.8 to 8.4], Standard Error of Mean 4.31
Statistical Analysis 7: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Role-Emotional; Test type: Superiority or Other; p = 0.7636, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-9.1 to 12.4], Standard Error of Mean 5.41
Statistical Analysis 8: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: SF-36 Mental Health Index; Test type: Superiority or Other; p = 0.7067, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 1.3, 95% CI 2-sided [-5.7 to 8.4], Standard Error of Mean 3.54
Statistical Analysis 9: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Physical Component Score; Test type: Superiority or Other; p = 0.8352, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-3.9 to 3.2], Standard Error of Mean 1.78
Statistical Analysis 10: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Mental Component Score; Test type: Superiority or Other; p = 0.9347, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-4.2 to 4.6], Standard Error of Mean 2.22

31. Secondary Outcome: Single-Blind Phase: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) at Week 6
Description: HADS: participant rated questionnaire with 2 subscales. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks); HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). Each subscale comprised of 7 items with range 0 (no presence of anxiety or depression) to 3 (severe feeling of anxiety or depression). Total score 0 to 21 for each subscale; higher score indicates greater severity of anxiety and depression symptoms.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  HADS-A Anxiety scale: number analyzed (Participants) | 421
  HADS-A Anxiety scale | -1.8 (3.47)
  HADS-D Depression scale: number analyzed (Participants) | 420
  HADS-D Depression scale | -1.5 (3.62)

32. Secondary Outcome: Double-Blind Phase: Change From Baseline in HADS Score at Week 19
Description: as for outcome 31
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  HADS-A Anxiety scale: number analyzed (Participants) | 60 | 57
  HADS-A Anxiety scale | -0.7 [-1.7 to 0.4] | -1.6 [-2.6 to -0.6]
  HADS-D Depression scale: number analyzed (Participants) | 60 | 57
  HADS-D Depression scale | -1.4 [-2.3 to -0.4] | -1.1 [-2.0 to -0.2]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); HADS-A Anxiety scale; Test type: Superiority or Other; p = 0.1901, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.9, 95% CI 2-sided [-0.5 to 2.3], Standard Error of Mean 0.69
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); HADS-D Depression scale; Test type: Superiority or Other; p = 0.6914, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.6 to 1.0], Standard Error of Mean 0.65

33. Secondary Outcome: Single-Blind Phase: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) at Week 6
Description: The FIQ is a 20-item self-administered questionnaire. FIQ contains 10 subscales, which are combined to yield a total score. There are 11 questions that are related specifically to physical functioning (item 1). The remaining questions assess pain, fatigue, stiffness, difficulty working, and symptoms of anxiousness and depression. The FIQ is scored from 0 to 100, with higher scores indicating more impairment.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  Item 1: Physical activities: number analyzed (Participants) | 288
  Item 1: Physical activities | -0.9 (2.14)
  Item 2: Feel good: number analyzed (Participants) | 288
  Item 2: Feel good | -2.2 (3.33)
  Item 3: Work missed: number analyzed (Participants) | 288
  Item 3: Work missed | -0.5 (2.42)
  Item 4: Do job: number analyzed (Participants) | 288
  Item 4: Do job | -1.5 (2.72)
  Item 5: Pain: number analyzed (Participants) | 288
  Item 5: Pain | -1.6 (2.25)
  Item 6: Fatigue: number analyzed (Participants) | 288
  Item 6: Fatigue | -1.4 (2.43)
  Item 7: Rested: number analyzed (Participants) | 288
  Item 7: Rested | -1.7 (2.65)
  Item 8: Stiffness: number analyzed (Participants) | 288
  Item 8: Stiffness | -1.8 (2.65)
  Item 9: Anxiety: number analyzed (Participants) | 288
  Item 9: Anxiety | -1.2 (2.95)
  Item 10: Depression: number analyzed (Participants) | 288
  Item 10: Depression | -0.6 (2.75)
  Total Score: number analyzed (Participants) | 288
  Total Score | -13.4 (16.71)

34. Secondary Outcome: Double-Blind Phase: Change From Baseline in FIQ Score at Week 19
Description: as for outcome 33
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Item 1: Physical activities: number analyzed (Participants) | 59 | 57
  Item 1: Physical activities | -1.0 [-1.6 to -0.4] | -1.3 [-1.9 to -0.8]
  Item 2: feel good: number analyzed (Participants) | 60 | 57
  Item 2: feel good | -3.0 [-3.9 to -2.1] | -3.2 [-4.1 to -2.3]
  Item 3: Work missed: number analyzed (Participants) | 60 | 57
  Item 3: Work missed | -1.2 [-1.7 to -0.7] | -1.0 [-1.5 to -0.5]
  Item 4: Do job: number analyzed (Participants) | 60 | 57
  Item 4: Do job | -2.1 [-3.0 to -1.3] | -2.2 [-3.0 to -1.4]
  Item 5: Pain: number analyzed (Participants) | 60 | 57
  Item 5: Pain | -2.7 [-3.4 to -2.0] | -2.2 [-2.8 to -1.5]
  Item 6: Fatigue: number analyzed (Participants) | 60 | 57
  Item 6: Fatigue | -2.3 [-3.0 to -1.6] | -2.4 [-3.0 to -1.7]
  Item 7: Rested: number analyzed (Participants) | 60 | 57
  Item 7: Rested | -2.6 [-3.4 to -1.8] | -2.2 [-3.0 to -1.4]
  Item 8: Stiffness: number analyzed (Participants) | 60 | 57
  Item 8: Stiffness | -2.4 [-3.2 to -1.6] | -2.2 [-3.0 to -1.4]
  Item 9: Anxiety: number analyzed (Participants) | 60 | 57
  Item 9: Anxiety | -1.8 [-2.6 to -1.0] | -1.7 [-2.5 to -0.9]
  Item 10: Depression: number analyzed (Participants) | 60 | 57
  Item 10: Depression | -0.7 [-1.4 to -0.0] | -0.7 [-1.3 to 0.0]
  Total Score: number analyzed (Participants) | 59 | 57
  Total Score | -19.6 [-25.3 to -13.9] | -19.1 [-24.6 to -13.7]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 1: Physical activities; Test type: Superiority or Other; p = 0.3721, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.5 to 1.2], Standard Error of Mean 0.41
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 2: Feel good; Test type: Superiority or Other; p = 0.8084, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-1.1 to 1.4], Standard Error of Mean 0.64
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 3: Work missed; Test type: Superiority or Other; p = 0.6312, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.9 to 0.5], Standard Error of Mean 0.35
Statistical Analysis 4: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 4: Do job; Test type: Superiority or Other; p = 0.8824, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-1.0 to 1.2], Standard Error of Mean 0.57
Statistical Analysis 5: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 5: Pain; Test type: Superiority or Other; p = 0.2742, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-1.5 to 0.4], Standard Error of Mean 0.49
Statistical Analysis 6: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 6: Fatigue; Test type: Superiority or Other; p = 0.8520, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.8 to 1.0], Standard Error of Mean 0.46
Statistical Analysis 7: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 7: Rested; Test type: Superiority or Other; p = 0.5264, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.4 to 0.7], Standard Error of Mean 0.55
Statistical Analysis 8: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 8: Stiffness; Test type: Superiority or Other; p = 0.6601, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.3 to 0.9], Standard Error of Mean 0.55
Statistical Analysis 9: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 9: Anxiety; Test type: Superiority or Other; p = 0.8937, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.2 to 1.0], Standard Error of Mean 0.56
Statistical Analysis 10: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Item 10: Depression; Test type: Superiority or Other; p = 0.9151, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-1.0 to 0.9], Standard Error of Mean 0.47
Statistical Analysis 11: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the total score; Test type: Superiority or Other; p = 0.9045, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-8.2 to 7.3], Standard Error of Mean 3.91

35. Secondary Outcome: Single-Blind Phase: Change From Baseline in Multidimensional Fatigue Inventory (MFI) at Week 6
Description: The MFI is a 20-item, self-administered questionnaire designed to measure the following dimensions of fatigue: general fatigue, physical fatigue, mental fatigue, reduced motivation, and reduced activity. Items are summed to form subscale scores; there is no overall score. The score range is from 4 to 20, where higher scores indicate greater dysfunction.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  General fatigue: number analyzed (Participants) | 289
  General fatigue | -0.2 (2.47)
  Physical fatigue: number analyzed (Participants) | 289
  Physical fatigue | 0.1 (2.67)
  Reduced activity: number analyzed (Participants) | 289
  Reduced activity | -0.2 (2.55)
  Reduced motivation: number analyzed (Participants) | 289
  Reduced motivation | 0.2 (2.71)
  Mental fatigue: number analyzed (Participants) | 289
  Mental fatigue | -0.1 (2.17)

36. Secondary Outcome: Double-Blind Phase: Change From Baseline in MFI Score at Week 19
Description: as for outcome 35
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  General fatigue: number analyzed (Participants) | 60 | 57
  General fatigue | 0.1 [-0.4 to 0.6] | -0.1 [-0.6 to 0.3]
  Physical fatigue: number analyzed (Participants) | 60 | 57
  Physical fatigue | -0.1 [-0.6 to 0.5] | 0.2 [-0.3 to 0.7]
  Reduced activity: number analyzed (Participants) | 60 | 57
  Reduced activity | 0.0 [-0.5 to 0.6] | -0.3 [-0.7 to 0.2]
  Reduced motivation: number analyzed (Participants) | 60 | 57
  Reduced motivation | 1.0 [0.4 to 1.5] | 0.3 [-0.2 to 0.8]
  Mental fatigue: number analyzed (Participants) | 60 | 57
  Mental fatigue | -0.1 [-0.5 to 0.3] | 0.1 [-0.3 to 0.4]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: General Fatigue; Test type: Superiority or Other; p = 0.4606, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.4 to 0.9], Standard Error of Mean 0.31
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Physical Fatigue; Test type: Superiority or Other; p = 0.4703, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-1.0 to 0.5], Standard Error of Mean 0.37
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Reduced activity; Test type: Superiority or Other; p = 0.4009, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.4 to 1.0], Standard Error of Mean 0.36
Statistical Analysis 4: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Reduced motivation; Test type: Superiority or Other; p = 0.0695, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.1 to 1.3], Standard Error of Mean 0.35
Statistical Analysis 5: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Mental fatigue; Test type: Superiority or Other; p = 0.5869, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.7 to 0.4], Standard Error of Mean 0.27

37. Secondary Outcome: Single-Blind Phase: Number of Participants With Benefit, Satisfaction, Willingness to Continue Measure (BSW) at Week 6
Description: The questionnaire consists of 3 single-item measures designed to captures the participant's perception of the effect of treatment in terms of the relative benefit, their satisfaction, and their intention or willingness to continue on therapy.
Time Frame: Week 6
Population: as for outcome 6
Measure: Number; unit: Participants
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Participants
  Benefit from treatment-No | 69
  Benefit from treatment-Little benefit | 137
  Benefit from treatment-much benefit | 211
  Satisfaction from treatment-very dissatisfied | 52
  Satisfaction from treatment-a little dissatisfied | 59
  Satisfaction from treatment-a little satisfied | 103
  Satisfaction from treatment-very satisfied | 203
  Willing to continue treatment-very unwilling | 68
  Willing to continue treatment-little unwilling | 33
  Willing to continue treatment-little bit willing | 49
  Willing to continue treatment-very willing | 266

38. Secondary Outcome: Double-Blind Phase: Number of Participants With Benefit, Satisfaction, and Willingness (BSW) to Continue Data at Visit 9 (3 Component Questions) at Week 19
Description: as for outcome 37
Time Frame: Week 19
Population: FAS consisted of all participants randomized to the DB phase who received at least 1 dose of study medication in the DB phase. Here, "overall number of participants analyzed" signifies participants evaluable for this outcome measure and "number analyzed"= participants evaluable for specified categories.
Measure: Number; unit: Participants
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 57
Participants
  Benefit from treatment-No: number analyzed (Participants) | 59 | 57
  Benefit from treatment-No | 3 | 11
  Benefit from treatment-Little benefit: number analyzed (Participants) | 59 | 57
  Benefit from treatment-Little benefit | 15 | 16
  Benefit from treatment-much benefit: number analyzed (Participants) | 59 | 57
  Benefit from treatment-much benefit | 41 | 30
  Satisfaction from treatment-very dissatisfied: number analyzed (Participants) | 60 | 57
  Satisfaction from treatment-very dissatisfied | 4 | 6
  Satisfaction from treatment-a little dissatisfied: number analyzed (Participants) | 60 | 57
  Satisfaction from treatment-a little dissatisfied | 10 | 8
  Satisfaction from treatment-a little satisfied: number analyzed (Participants) | 60 | 57
  Satisfaction from treatment-a little satisfied | 10 | 13
  Satisfaction from treatment-very satisfied: number analyzed (Participants) | 60 | 57
  Satisfaction from treatment-very satisfied | 36 | 30
  Willing to continue treatment-very unwilling: number analyzed (Participants) | 60 | 57
  Willing to continue treatment-very unwilling | 8 | 4
  Willing to continue treatment-little unwilling: number analyzed (Participants) | 60 | 57
  Willing to continue treatment-little unwilling | 6 | 8
  Willing to continue treatment-little bit willing: number analyzed (Participants) | 60 | 57
  Willing to continue treatment-little bit willing | 9 | 11
  Willing to continue treatment-very willing: number analyzed (Participants) | 60 | 57
  Willing to continue treatment-very willing | 37 | 34
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Benefit from treatment; Test type: Superiority or Other; p = 0.0296, two-sided test — Nominal p-value for two-sided test; Odds Ratio (OR) = 2.29, 95% CI 2-sided [1.09 to 4.81]
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Satisfaction from treatment; Test type: Superiority or Other; p = 0.4691, two-sided test — Nominal p-value for two-sided test; Odds Ratio (OR) = 1.29, 95% CI 2-sided [0.64 to 2.61]
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Willingness to continue treatment; Test type: Superiority or Other; p = 0.9577, two-sided test — Nominal p-value for two-sided test; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.48 to 2.01]

39. Secondary Outcome: Single-Blind Phase: Change From Baseline in Work Productivity and Activity Impairment (WPAI) Questionnaire at Week 6
Description: WPAI: 6 question participant rated questionnaire to determine the degree to which disease state affected work productivity while at work and affected activities outside of work. Subscale scores include percent work time missed due to the health problem; percent impairment while working due to problem; percent overall work impairment due to problem; and percent activity impairment due to problem. Scores scaled as 0 (not affected/no impairment) to 10 (completely affected/impaired). Higher scores indicated greater impairment and less productivity.
Time Frame: Baseline, Week 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Units on a scale
  Percent Work Time Missed: number analyzed (Participants) | 134
  Percent Work Time Missed | -5.8 (48.69)
  Percent Impairment While Working: number analyzed (Participants) | 109
  Percent Impairment While Working | -10.0 (31.29)
  Percent Activity Impairment: number analyzed (Participants) | 272
  Percent Activity Impairment | -13.5 (25.88)
  Percent Overall Work Impairment: number analyzed (Participants) | 274
  Percent Overall Work Impairment | -12.3 (27.62)

40. Secondary Outcome: Double-Blind Phase: Change From Baseline WPAI Questionnaire at Week 19
Description: as for outcome 39
Time Frame: Baseline, Week 19
Population: as for outcome 7
Measure: Least Squares Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Units on a scale
  Percent Work Time Missed: number analyzed (Participants) | 31 | 30
  Percent Work Time Missed | -7.3 [-21.3 to 6.7] | -26.7 [-41.0 to -12.3]
  Percent Impairment While Working: number analyzed (Participants) | 24 | 24
  Percent Impairment While Working | -14.0 [-19.7 to -8.2] | -15.0 [-20.8 to -9.3]
  Percent Activity Impairment: number analyzed (Participants) | 56 | 52
  Percent Activity Impairment | -16.4 [-19.0 to -13.7] | -19.6 [-22.1 to -17.0]
  Percent Overall Work Impairment: number analyzed (Participants) | 56 | 52
  Percent Overall Work Impairment | -15.9 [-18.7 to -13.1] | -17.5 [-20.2 to -14.8]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Percent Work Time Missed; Test type: Superiority or Other; p = 0.0562, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 19.3, 95% CI 2-sided [-0.5 to 39.2], Standard Error of Mean 9.85
Statistical Analysis 2: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Percent Impairment While Working; Test type: Superiority or Other; p = 0.7892, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 1.1, 95% CI 2-sided [-7.0 to 9.2], Standard Error of Mean 3.96
Statistical Analysis 3: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Percent Activity Impairment; Test type: Superiority or Other; p = 0.0819, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 3.2, 95% CI 2-sided [-0.4 to 6.8], Standard Error of Mean 1.82
Statistical Analysis 4: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Percent Overall Work Impairment; Test type: Superiority or Other; p = 0.4135, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 1.6, 95% CI 2-sided [-2.2 to 5.4], Standard Error of Mean 1.91

41. Other Pre Specified Outcome: Single-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Total Sleep Time at Weeks 3, 4, 5, 6 and 7
Description: Actigraphy was assessed with an accelerometer that was worn on the wrist. The accelerometer was programmed to record movements. This information was used to calculate several endpoints reflecting daytime activity, and sleep quality and duration. Total sleep time = number of minutes asleep between time of sleep onset to morning awakening.
Time Frame: Baseline, Weeks 3, 4, 5, 6 and 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Hours
  Total Sleep Time (Week 3): number analyzed (Participants) | 16
  Total Sleep Time (Week 3) | -0.1 (0.94)
  Total Sleep Time (Week 4): number analyzed (Participants) | 302
  Total Sleep Time (Week 4) | 0.4 (0.99)
  Total Sleep Time (Week 5): number analyzed (Participants) | 292
  Total Sleep Time (Week 5) | 0.3 (1.02)
  Total Sleep Time (Week 6): number analyzed (Participants) | 211
  Total Sleep Time (Week 6) | 0.3 (1.15)
  Total Sleep Time (Week 7): number analyzed (Participants) | 10
  Total Sleep Time (Week 7) | 0.6 (1.10)

42. Other Pre Specified Outcome: Single-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Minutes of Interrupted Sleep at Weeks 3, 4, 5, 6 and 7
Description: Actigraphy was assessed with an accelerometer that was worn on the wrist. The accelerometer was programmed to record movements. This information was used to calculate several endpoints reflecting daytime activity, and sleep quality and duration. Minutes of interrupted sleep = minutes awake after sleep onset (analogous to wake-time after sleep onset from polysomnography measurements).
Time Frame: Baseline, Weeks 3, 4, 5, 6 and 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Minutes
  Minutes of Interrupted Sleep (Week 3): number analyzed (Participants) | 16
  Minutes of Interrupted Sleep (Week 3) | -5.3 (12.63)
  Minutes of Interrupted Sleep (Week 4): number analyzed (Participants) | 302
  Minutes of Interrupted Sleep (Week 4) | -5.9 (16.10)
  Minutes of Interrupted Sleep (Week 5): number analyzed (Participants) | 292
  Minutes of Interrupted Sleep (Week 5) | -7.0 (15.66)
  Minutes of Interrupted Sleep (Week 6): number analyzed (Participants) | 211
  Minutes of Interrupted Sleep (Week 6) | -6.6 (16.12)
  Minutes of Interrupted Sleep (Week 7): number analyzed (Participants) | 10
  Minutes of Interrupted Sleep (Week 7) | 0.7 (19.43)

43. Other Pre Specified Outcome: Single-Blind Phase: Change From Baseline at in Actigraphy Functional/Sleep Assessment - Sleep Fragmentation Index Weeks 3, 4, 5, 6 and 7
Description: Actigraphy was assessed with an accelerometer that was worn on the wrist. The accelerometer was programmed to record movements. This information was used to calculate several endpoints reflecting daytime activity, and sleep quality and duration. Sleep fragmentation index = a measure of sleep relatedness. Sleep fragmentation index calculated from analysis of the periods that participant was not moving (immobile bouts). It is number of immobile bouts that were exactly 1 minute long divided by total number of immobile bouts. Value ranges from 0-100 percent, with low number representing more restful sleep.
Time Frame: Baseline, Weeks 3, 4, 5, 6 and 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percentage of immobile bouts
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Percentage of immobile bouts
  Sleep Fragmentation Index (Week 3): number analyzed (Participants) | 16
  Sleep Fragmentation Index (Week 3) | -0.8 (5.27)
  Sleep Fragmentation Index (Week 4): number analyzed (Participants) | 302
  Sleep Fragmentation Index (Week 4) | -2.5 (5.45)
  Sleep Fragmentation Index (Week 5): number analyzed (Participants) | 292
  Sleep Fragmentation Index (Week 5) | -2.8 (5.27)
  Sleep Fragmentation Index (Week 6): number analyzed (Participants) | 211
  Sleep Fragmentation Index (Week 6) | -2.6 (5.63)
  Sleep Fragmentation Index (Week 7): number analyzed (Participants) | 10
  Sleep Fragmentation Index (Week 7) | 0.7 (5.85)

44. Other Pre Specified Outcome: Single-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Total Daytime Activity at Weeks 3, 4, 5, 6 and 7
Description: Actigraphy was assessed with an accelerometer that was worn on the wrist. The accelerometer was programmed to record movements. This information was used to calculate several endpoints reflecting daytime activity, and sleep quality and duration. Total daytime activity = total activity "counts" during the day.
Time Frame: Baseline, Weeks 3, 4, 5, 6 and 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Counts of total daytime activity
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Counts of total daytime activity
  Total daytime activity (Week 3): number analyzed (Participants) | 16
  Total daytime activity (Week 3) | 10264.3 (90090.07)
  Total daytime activity (Week 4): number analyzed (Participants) | 297
  Total daytime activity (Week 4) | 10588.1 (59150.38)
  Total daytime activity (Week 5): number analyzed (Participants) | 287
  Total daytime activity (Week 5) | 8635.8 (54823.64)
  Total daytime activity (Week 6): number analyzed (Participants) | 208
  Total daytime activity (Week 6) | 7134.2 (58221.22)
  Total daytime activity (Week 7): number analyzed (Participants) | 10
  Total daytime activity (Week 7) | 18420.7 (61725.84)

45. Other Pre Specified Outcome: Single-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Percent Sedentary at Weeks 3, 4, 5, 6 and 7
Description: Actigraphy was assessed with an accelerometer that was worn on the wrist. The accelerometer was programmed to record movements. This information was used to calculate several endpoints reflecting daytime activity, and sleep quality and duration. Percent sedentary = percent of daytime spent in sedentary activities as determined by the activity counts measured each minute.
Time Frame: Baseline, Weeks 3, 4, 5, 6 and 7
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Percent of daytime
Arm/Group | Pregabalin (Single Blind Phase)
Number analyzed (Participants) | 441
Percent of daytime
  Percent Sedentary (Week 3): number analyzed (Participants) | 16
  Percent Sedentary (Week 3) | 0.7 (6.66)
  Percent Sedentary (Week 4): number analyzed (Participants) | 302
  Percent Sedentary (Week 4) | 0.7 (5.61)
  Percent Sedentary (Week 5): number analyzed (Participants) | 292
  Percent Sedentary (Week 5) | 0.6 (5.62)
  Percent Sedentary (Week 6): number analyzed (Participants) | 211
  Percent Sedentary (Week 6) | 0.3 (6.07)
  Percent Sedentary (Week 7): number analyzed (Participants) | 10
  Percent Sedentary (Week 7) | 0.2 (5.51)

46. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Total Sleep Time at Weeks 11, 12, 13, 14 and 15
Description: as for outcome 41
Time Frame: Baseline, Weeks 11, 12, 13, 14 and 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Hours
  Total Sleep Time (Week 11): number analyzed (Participants) | 9 | 12
  Total Sleep Time (Week 11) | 0.5 (0.91) | 0.0 (1.53)
  Total Sleep Time (Week 12): number analyzed (Participants) | 43 | 37
  Total Sleep Time (Week 12) | 0.5 (1.23) | 0.1 (1.01)
  Total Sleep Time (Week 13): number analyzed (Participants) | 40 | 36
  Total Sleep Time (Week 13) | 0.4 (1.15) | 0.1 (1.15)
  Total Sleep Time (Week 14): number analyzed (Participants) | 37 | 36
  Total Sleep Time (Week 14) | 0.4 (1.02) | 0.1 (1.14)
  Total Sleep Time (Week 15): number analyzed (Participants) | 22 | 17
  Total Sleep Time (Week 15) | 0.2 (0.91) | 0.3 (1.13)

47. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Minutes of Interrupted Sleep at Weeks 11, 12, 13, 14 and 15
Description: as for outcome 42
Time Frame: Baseline, Weeks 11, 12, 13, 14 and 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Minutes
  Minutes of Interrupted Sleep (Week 11): number analyzed (Participants) | 9 | 12
  Minutes of Interrupted Sleep (Week 11) | -9.0 (10.27) | 2.5 (18.97)
  Minutes of Interrupted Sleep (Week 12): number analyzed (Participants) | 43 | 37
  Minutes of Interrupted Sleep (Week 12) | -3.0 (14.77) | -1.7 (14.10)
  Minutes of Interrupted Sleep (Week 13): number analyzed (Participants) | 40 | 36
  Minutes of Interrupted Sleep (Week 13) | -3.0 (20.33) | 0.4 (14.14)
  Minutes of Interrupted Sleep (Week 14): number analyzed (Participants) | 37 | 36
  Minutes of Interrupted Sleep (Week 14) | -3.2 (19.12) | -1.8 (13.19)
  Minutes of Interrupted Sleep (Week 15): number analyzed (Participants) | 22 | 17
  Minutes of Interrupted Sleep (Week 15) | -0.4 (25.03) | -0.5 (13.73)

48. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Sleep Fragmentation Index at Weeks 11, 12, 13, 14 and 15
Description: as for outcome 43
Time Frame: Baseline, Weeks 11, 12, 13, 14 and 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percentage of immobile bouts
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Percentage of immobile bouts
  Sleep Fragmentation Index (Week 11): number analyzed (Participants) | 9 | 12
  Sleep Fragmentation Index (Week 11) | -4.4 (5.53) | 0.1 (5.17)
  Sleep Fragmentation Index (Week 12): number analyzed (Participants) | 43 | 37
  Sleep Fragmentation Index (Week 12) | -2.8 (5.91) | -0.4 (6.29)
  Sleep Fragmentation Index (Week 13): number analyzed (Participants) | 40 | 36
  Sleep Fragmentation Index (Week 13) | -2.2 (7.28) | -0.3 (5.23)
  Sleep Fragmentation Index (Week 14): number analyzed (Participants) | 37 | 36
  Sleep Fragmentation Index (Week 14) | -2.4 (7.32) | -0.6 (4.75)
  Sleep Fragmentation Index (Week 15): number analyzed (Participants) | 22 | 17
  Sleep Fragmentation Index (Week 15) | -0.9 (7.41) | -0.9 (5.19)

49. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Total Daytime Activity at Weeks 11, 12, 13, 14 and 15
Description: as for outcome 44
Time Frame: Baseline, Weeks 11, 12, 13, 14 and 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Counts of total daytime activity
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Counts of total daytime activity
  Total daytime activity (Week 11): number analyzed (Participants) | 9 | 12
  Total daytime activity (Week 11) | -1894.1 (46879.81) | -2083.9 (40939.67)
  Total daytime activity ((Week 12): number analyzed (Participants) | 43 | 37
  Total daytime activity ((Week 12) | -50.7 (50114.87) | -6691.1 (47353.03)
  Total daytime activity ((Week 13): number analyzed (Participants) | 40 | 36
  Total daytime activity ((Week 13) | -4362.4 (51922.75) | 521.8 (46996.71)
  Total daytime activity ((Week 14): number analyzed (Participants) | 37 | 36
  Total daytime activity ((Week 14) | -179.7 (55858.35) | -4523.8 (52629.95)
  Total daytime activity ((Week 15): number analyzed (Participants) | 22 | 17
  Total daytime activity ((Week 15) | -4138.3 (54924.02) | -4649.4 (58121.16)

50. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Percent Sedentary at Weeks 11, 12, 13, 14 and 15
Description: as for outcome 45
Time Frame: Baseline, Weeks 11, 12, 13, 14 and 15
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Percent of daytime
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 63 | 58
Percent of daytime
  Percent Sedentary (Week 11): number analyzed (Participants) | 9 | 12
  Percent Sedentary (Week 11) | -0.7 (7.72) | 1.1 (6.69)
  Percent Sedentary (Week 12): number analyzed (Participants) | 43 | 37
  Percent Sedentary (Week 12) | -0.8 (5.66) | -1.4 (6.15)
  Percent Sedentary (Week 13): number analyzed (Participants) | 40 | 36
  Percent Sedentary (Week 13) | -1.3 (5.41) | -0.9 (6.15)
  Percent Sedentary (Week 14): number analyzed (Participants) | 37 | 36
  Percent Sedentary (Week 14) | -2.1 (6.56) | -1.1 (7.27)
  Percent Sedentary (Week 15): number analyzed (Participants) | 22 | 17
  Percent Sedentary (Week 15) | -1.5 (5.21) | -1.4 (6.56)

51. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment- Total Sleep Time at Double Blind End Point Visit (Week 19)
Description: as for outcome 41
Time Frame: Baseline, Double blind end point visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Hours
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 44 | 38
Hours | 0.5 [0.1 to 0.9] | 0.1 [-0.3 to 0.5]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.1224, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.1 to 0.9], Standard Error of Mean 0.24

52. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Minutes of Interrupted Sleep at Double Blind End Point Visit (Week 19)
Description: as for outcome 42
Time Frame: Baseline, Double blind end point visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Minutes
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 44 | 38
Minutes | -3.5 [-10.0 to 2.9] | -2.3 [-8.8 to 4.1]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.7680, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-9.3 to 6.9], Standard Error of Mean 4.06

53. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Sleep Fragmentation Index at Double Blind End Point Visit (Week 19)
Description: as for outcome 43
Time Frame: Baseline, Double blind end point visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of immobile bouts
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 44 | 38
Percentage of immobile bouts | -2.5 [-4.6 to -0.5] | -0.6 [-2.6 to 1.4]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.1360, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = -1.9, 95% CI 2-sided [-4.5 to 0.6], Standard Error of Mean 1.29

54. Secondary Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Total Daytime Activity at Double Blind End Point Visit (Week 19)
Description: as for outcome 44
Time Frame: Baseline, Double blind end point visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Counts of total daytime activity
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 44 | 38
Counts of total daytime activity | -182.7 [-20143.1 to 19777.7] | -6672.2 [-26663.5 to 13319.1]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); This analysis is for the domain: Total daytime activity; Test type: Superiority or Other; p = 0.6077, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 6489.5, 95% CI 2-sided [-18648.6 to 31627.6], Standard Error of Mean 12579.50

55. Other Pre Specified Outcome: Double-Blind Phase: Change From Baseline in Actigraphy Functional/Sleep Assessment - Percent Sedentary at Double Blind End Point Visit (Week 19)
Description: as for outcome 45
Time Frame: Baseline, Double blind end point visit (Week 19)
Population: as for outcome 5
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent of daytime
Arm/Group | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 44 | 38
Percent of daytime | -1.4 [-3.6 to 0.8] | -2.0 [-4.2 to 0.2]
Statistical Analysis 1: Comparison: Pregabalin (Double Blind Phase) vs Placebo (Double Blind Phase); Test type: Superiority or Other; p = 0.6647, ANCOVA — Estimates and p-values are from a ANCOVA main effects model with baseline value, center, treatment in the model; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-2.2 to 3.4], Standard Error of Mean 1.38

56. Other Pre Specified Outcome: Number of Participants With Suicidal Ideation Throughout the Study Assessed by Columbia Classification Algorithm of Suicide Assessment (C-CASA)
Description: C-CASA was used to categorize and summarize results from the Sheehan Suicidality Tracking Scale (S-STS) and the Columbia Suicidality Severity Rating Scale (C-SSRS). S-STS was an 8-item prospective rating scale that tracked treatment-emergent suicidal ideation and behaviors. Items 1a, 2 to 6, 7a, 8 were scored on a 5-point Likert scale (ranges 0 [not at all] to 4 [extremely]). Items 1, 1b, and 7 required yes or no responses. S-STS total score range 0-30. Lower score=reduced suicidal tendency. C-SSRS was a participant rated questionnaire to assess suicidal ideation, suicidal behavior, actual attempts (yes or no responses), and intensity of ideation (rated 1=low severity to 5=high severity). Responses on S-STS or C-SSRS were mapped to C-CASA categories as: Completed suicide; suicide attempt; preparatory acts; suicide ideation; self-injurious behavior, intent unknown; not enough information; self-injurious behavior, no suicide intent; other, no deliberate self harm.
Time Frame: Week 1 to Week 7 and Week 11 to Week 20
Population: The population in the single and double blind phase consisted of all paticipants who received at least 1 dose of study medication and who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Pregabalin (Single Blind Phase) | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Number analyzed (Participants) | 441 | 63 | 58
Participants
  Week 1: number analyzed (Participants) | 426 | 0 | 0
  Week 1 | 5 |  |
  Week 2: number analyzed (Participants) | 408 | 0 | 0
  Week 2 | 6 |  |
  Week 3: number analyzed (Participants) | 381 | 0 | 0
  Week 3 | 4 |  |
  Week 6: number analyzed (Participants) | 422 | 0 | 0
  Week 6 | 16 |  |
  Week 7: number analyzed (Participants) | 273 | 0 | 0
  Week 7 | 10 |  |
  Week 11: number analyzed (Participants) | 0 | 55 | 50
  Week 11 |  | 3 | 0
  Week 15: number analyzed (Participants) | 0 | 49 | 47
  Week 15 |  | 1 | 1
  Week 19: number analyzed (Participants) | 0 | 60 | 57
  Week 19 |  | 1 | 3
  Week 20: number analyzed (Participants) | 0 | 56 | 52
  Week 20 |  | 1 | 1

ADVERSE EVENTS:
Time Frame: From time that the participant provided informed consent through and including 28 calender days after the last administration of the investigational product (up to Week 20)
Description: The same event may appear as both an AE and a serious AE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Pregabalin (Single Blind Phase) | Pregabalin (Double Blind Phase) | Placebo (Double Blind Phase)
Serious Adverse Events (participants affected / at risk) | 5/441 | 2/63 | 0/58
Other Adverse Events (participants affected / at risk) | 353/441 | 34/63 | 27/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (Single Blind Phase) (N=441) | Pregabalin (Double Blind Phase) (N=63) | Placebo (Double Blind Phase) (N=58)
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Hypertension (Investigations) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (Single Blind Phase) (N=441) | Pregabalin (Double Blind Phase) (N=63) | Placebo (Double Blind Phase) (N=58)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 5 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 1 | 0
Dry eye (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 1 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Keratitis (Eye disorders) | 1 | 0 | 0
Diplopia (Eye disorders) | 2 | 0 | 0
Vision blurred (Eye disorders) | 29 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0
Visual impairment (Eye disorders) | 2 | 0 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0
Gingival disorder (Gastrointestinal disorders) | 1 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 1 | 0
Gastric disorder (Gastrointestinal disorders) | 1 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 19 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 13 | 1 | 2
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 6 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 9 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 6 | 0 | 0
Mucous stools (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 41 | 5 | 0
Vomiting (Gastrointestinal disorders) | 12 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 25 | 0 | 2
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 4 | 0 | 0
Chest discomfort (General disorders) | 2 | 0 | 2
Chest pain (General disorders) | 4 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Face oedema (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 42 | 1 | 0
Feeling abnormal (General disorders) | 17 | 2 | 0
Feeling drunk (General disorders) | 3 | 0 | 0
Feeling hot (General disorders) | 2 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
Generalised oedema (General disorders) | 2 | 1 | 0
Gravitational oedema (General disorders) | 1 | 0 | 0
Irritability (Psychiatric disorders) | 4 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Mucosal dryness (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0
Oedema (General disorders) | 5 | 0 | 0
Oedema peripheral (General disorders) | 27 | 6 | 2
Pain (General disorders) | 3 | 0 | 0
Sluggishness (General disorders) | 1 | 0 | 0
Swelling (General disorders) | 3 | 0 | 0
Thirst (General disorders) | 2 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Pertussis (Infections and infestations) | 1 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 1 | 0
Tinea pedis (Infections and infestations) | 0 | 1 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 5 | 0 | 1
Cystitis (Infections and infestations) | 2 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Kidney infection (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1 | 3
Otitis media (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 11 | 1 | 1
Urinary tract infection (Infections and infestations) | 12 | 1 | 1
Vulvovaginitis (Infections and infestations) | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 2 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 2 | 0 | 0
Bone contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 2 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 2 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood pressure diastolic increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 3 | 1 | 0
Cardiac murmur (Investigations) | 0 | 1 | 0
Heart sounds abnormal (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood glucose increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0
Bacterial test positive (Investigations) | 1 | 0 | 0
Helicobacter test positive (Investigations) | 1 | 0 | 0
Neurological examination abnormal (Investigations) | 1 | 0 | 0
Weight increased (Investigations) | 30 | 2 | 1
Glucose urine present (Investigations) | 1 | 0 | 0
Blood calcium decreased (Investigations) | 1 | 0 | 0
Blood potassium increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Food craving (Metabolism and nutrition disorders) | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 20 | 0 | 0
Fluid retention (Metabolism and nutrition disorders) | 2 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 8 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 12 | 0 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myokymia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 43 | 1 | 2
Migraine (Nervous system disorders) | 0 | 1 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0
Amnesia (Nervous system disorders) | 3 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Disturbance in attention (Nervous system disorders) | 24 | 0 | 0
Memory impairment (Nervous system disorders) | 6 | 2 | 0
Mental impairment (Nervous system disorders) | 9 | 0 | 0
Bradykinesia (Nervous system disorders) | 1 | 0 | 0
Dyskinesia (Nervous system disorders) | 1 | 0 | 0
Psychomotor hyperactivity (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 5 | 0 | 0
Ataxia (Nervous system disorders) | 3 | 0 | 0
Balance disorder (Nervous system disorders) | 19 | 0 | 0
Coordination abnormal (Nervous system disorders) | 6 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 161 | 2 | 2
Dysarthria (Nervous system disorders) | 4 | 0 | 0
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Lethargy (Nervous system disorders) | 2 | 0 | 0
Paraesthesia (Nervous system disorders) | 4 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Sedation (Nervous system disorders) | 11 | 0 | 0
Sensory disturbance (Nervous system disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 105 | 0 | 0
Hypersomnia (Nervous system disorders) | 4 | 0 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0 | 0
Acute stress disorder (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 6 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 1 | 0 | 0
Generalised anxiety disorder (Psychiatric disorders) | 0 | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0 | 0
Stress (Psychiatric disorders) | 2 | 0 | 0
Attention deficit/hyperactivity disorder (Psychiatric disorders) | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 6 | 1 | 0
Disorientation (Psychiatric disorders) | 3 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 1
Depression (Psychiatric disorders) | 4 | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0 | 0
Bradyphrenia (Psychiatric disorders) | 2 | 0 | 0
Bipolar II disorder (Psychiatric disorders) | 1 | 0 | 0
Affect lability (Psychiatric disorders) | 2 | 0 | 1
Dysphoria (Psychiatric disorders) | 1 | 0 | 0
Emotional disorder (Psychiatric disorders) | 1 | 0 | 0
Euphoric mood (Psychiatric disorders) | 10 | 0 | 0
Mood swings (Psychiatric disorders) | 0 | 1 | 0
Aggression (Psychiatric disorders) | 2 | 0 | 0
Psychiatric symptom (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 2 | 0 | 0
Anorgasmia (Psychiatric disorders) | 1 | 0 | 0
Libido decreased (Psychiatric disorders) | 3 | 0 | 0
Abnormal dreams (Psychiatric disorders) | 2 | 0 | 0
Initial insomnia (Psychiatric disorders) | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 24 | 3 | 1
Nightmare (Psychiatric disorders) | 2 | 0 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0 | 1
Somnambulism (Psychiatric disorders) | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1
Enuresis (Renal and urinary disorders) | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 3 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 3 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 1
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Snoring (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 5 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Skin warm (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Raynaud's phenomenon (Vascular disorders) | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 1 | 0
Hot flush (Vascular disorders) | 2 | 1 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 10 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Post-traumatic stress disorder (Psychiatric disorders) | 1 | 0 | 0
Peripheral venous disease (Vascular disorders) | 1 | 0 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.